CLINICAL TRIAL: NCT03686163
Title: Effects of Intranasal Nerve Growth Factor for Acute Ischemic Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Xinfeng Liu, Professor, Jinling Hospital, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NGF-ischemic stroke
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic stroke; Nerve Growth Factor; Intranasal; Neurological Function
MeSH Terms: conditions — Ischemic Stroke; Hereditary Sensory and Autonomic Neuropathies | interventions — Nerve Growth Factors; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IN-NGF group (Experimental): Patients who underwent acute ischemic stroke will be chosen to receive NGF randomly
  Interventions: Drug: Nerve Growth Factors
- Control group (Placebo Comparator): Patients who underwent acute ischemic stroke will be chosen to receive normal saline randomly
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Nerve Growth Factors — the experimental group patients will receive NGF 20ug/d intranasally for 2 weeks
  Arms: IN-NGF group
Drug: normal saline — The Placebo Comparator group patients will receive nomral saline 20ug/d intranasally for 2 weeks
  Arms: Control group

SUMMARY:
Stroke remains one of the leading causes of death and adult disability worldwide. Yet, currently, the only accepted treatment for acute ischemic stroke(AIS) is recanalization of occluded arteries. Thrombolysis with tissue plasminogen activator, limited by its narrow therapeutic time window and the concern of hemorrhagic complication, is still uncommon in use. The other approach is to try to impede the ischemic cascade by targeting various components of the cascade that are deemed to be of importance, namely, a neuroprotection strategy.

Nerve growth factor (NGF) plays extensive roles in preventing ischemic injury. Besides that, it is also involved in neurogenesis of the central nervous system (CNS). In addition, the levels of NGF protein and messenger RNA significantly decreased in the CNS at the first few hours and returned to normal levels several days later after middle cerebral artery occlusion (MCAO) in animal models. These observed results suggested that NGF was demanded in ischemic brain injury, but endogenous NGF is insufficient for the requirement and delivering exogenous ones will be blocked in entering into the CNS by the blood-brain barrier (BBB). Intracerebroventricular or intracerebral injection of NGF or grafting of NGF-producing cells may be less practicable due to invasiveness and safety concerns.

Intranasal (IN) administration is a noninvasive and acceptable delivery strategy for drugs bypassing BBB and can deliver NGF to the CNS, which has been proved to show neuroprotective effects on brain injury.

The effects of intranasal NGF in human ischemic stroke is still controversial that need further evaluation.

DETAILED DESCRIPTION:
The proposed study is a randomized, double-blind, placebo-controlled trail of NGF, starting between 24 to 72 hours post acute ischemic stroke, continuing for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18years;
2. Acute ischemic stroke consistent within 72 hours;
3. Written informed consent from patient or surrogate, if unable to provide consent.

Exclusion Criteria:

1. Premorbid mRS ≥ 3 points;
2. Currently in pregnant or lactating;
3. Allergy to NGF;
4. Current participation in another investigation drug or device study;
5. Life expectancy less than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
a favorable neurological function | at 90 days post-treatment
  The primary outcome is determined as a favorable neurological function which is defined as Modified Rankin Scale(mRS) score of 0-3

CONTACTS AND LOCATIONS:
Overall Officials: Xinfeng Liu, MD, Study Chair — Department of Neurology, Jinling Hospital, China
Locations (1):
- Department of Neurology, Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No